CLINICAL TRIAL: NCT04042818
Title: Reliability of Rehabilitative Ultrasound Imaging for the Quadriceps Muscle and Sarcopenia in Poststroke Patients
Brief Title: Reliability of Rehabilitative Ultrasound for the Quadriceps Muscle and Sarcopenia in Poststroke Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Akif GÜLER, Principal Investigator, Gaziosmanpasa Research and Education Hospital
Other Study IDs: GaziosmanpasaTREH7
Record Dates: First submitted 2019-07-20; First posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Sarcopenia; Stroke, Complication; Quadriceps Muscle Atrophy; Hemiplegia; Ultrasonography; Hand Strength
Keywords: Sarcopenia; Stroke; Quadriceps Muscle Atrophy; Hemiplegia; Ultrasonography; Hand Strength
MeSH Terms: conditions — Sarcopenia; Stroke; Hemiplegia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Rehabilitative Ultrasound — Ultrasound imagining

SUMMARY:
The purpose of the study is search the interrater and intrarater reliability of the quadriceps muscle using rehabilitative ultrasound imaging and search for an association between sarcopenia and quadriceps muscle in poststroke patients.

DETAILED DESCRIPTION:
Poststroke patients often suffer from muscle atrophy in quadriceps muscle. Quadriceps muscle is essential for independent standing or ambulation after stroke. Quadriceps muscle consists of four different muscles: rectus femoris, vastus intermedius, vastus lateralis and medialis. The present study search for reliability for rectus femoris and vastus intermedius muscle thickness and cross-sectional area using rehabilitative ultrasound imagining. Longitudinal and transverse ultrasound imagining of the muscle thickness will be performed on both rectus femoris and vastus intermedius muscles for both extremities. The procedures will be repeated by two experts at two separate times (7-10 days). For sarcopenia measurement grip strength and DEXA measurements of the patients will be calculated. Totally 68 patients will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Poststroke patients (>6 months)

Exclusion Criteria:

* < 6 months after stroke
* Multiple stroke

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Poststroke patients
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
Thickness of Rectus Femoris Muscle | One week
  Longitudinal and Transverse thickness of rectus femoris muscle
Thickness of vastus intermedius muscle | One week
  Longitudinal and Transverse thickness of vastus intermedius muscle
Cross-sectional area of Rectus Femoris Muscle | One week
  Cross-sectional area of Rectus Femoris Muscle

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Y Yalçınkaya, M.D., Study Director — Gaziosmanpasa Taksim Training and Research Hospital
Locations (1):
- Gaziosmanpasa Taksim Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No